CLINICAL TRIAL: NCT07264231
Title: Benefits of Exercise for the Maternal-Fetal Unit During Pregnancy
Brief Title: Exercise During Pregnancy: Effects on the Maternal-Fetal Unit
Acronym: PREGFIT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Pública de Navarra (Other)
Collaborators: Instituto de Investigación Sanitaria de Navarra (IdiSNA) (Unknown); NavarraBiomed Biomedical Research Center (Other); Complejo Hospitalario de Navarra (Other)
Responsible Party: Principal Investigator, Robinson Ramírez-Vélez, Principal Investigator, Universidad Pública de Navarra
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PI_2024/148
Record Dates: First submitted 2025-09-23; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Pregnancy
Keywords: Exercise; Motor Activity
MeSH Terms: conditions — Motor Activity | interventions — Methods

STUDY DESIGN:
Intervention Model Description: Supervised exercise training: the women will attend at least 2 weekly sessions consisting of aerobic exercise (walking on treadmills), strength training (for upper body, back, abdomen and legs) as well as pelvic floor muscle exercises. Each session is 60 minutes and lead by a exercise physiologist. The women will also go through motivational interviewing sessions throughout the intervention period and are encouraged to do home exercise training in addition to the supervised exercise.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise training (Experimental): Participants will perform a supervised aerobic exercise program at 70% of maximum heart rate (HRmax), for 45 minutes per session, 3 times per week, during 12 weeks. Each session will follow a standardized protocol: 10 minutes of warm-up, 30 minutes of aerobic exercise, 5 minutes of cool-down and stretching. In addition, strength training sessions will be included 1-2 times per week.
  All exercise sessions will be delivered by qualified professionals, including exercise specialists, nutritionists, and physiotherapists with >3 years of experience and a master's-level education in the field. The intervention will be conducted at the Exercise Physiology Unit (E-FIT Group Laboratory), Navarrabiomed Research Center, Pamplona, Spain.
  Interventions: Behavioral: Intervention
- Control (No Intervention): Usual care as provided by the health services in Spain. The investigators will not advice the women to be inactive.

INTERVENTIONS:
Behavioral: Intervention — Exercise
  Arms: Exercise training

SUMMARY:
Metabolic alterations during pregnancy have been associated with adverse maternal-fetal outcomes, including low birth weight and pregnancy complications. Maternal endothelial dysfunction, oxidative stress, insulin resistance, and placental mitochondrial dysfunction are thought to contribute to fetal metabolic disturbances. Lifestyle changes, such as structured exercise during pregnancy, may modulate maternal and placental factors.

This randomized controlled trial will evaluate the effects of a multicomponent exercise program during the second and third trimester on maternal functional capacity, vascular health, anthropometry, metabolic biomarkers, placental function, and newborn health outcomes.

DETAILED DESCRIPTION:
To investigate the effects of a multicomponent supervised exercise program during pregnancy on the maternal-fetal unit.

ELIGIBILITY:
Inclusion Criteria:

* Primigravid women
* Gestational age 16-20 weeks
* No severe malformations on ultrasound
* Regular prenatal care and medical clearance from obstetrician
* Being healthy and able to exercise following American College of Obstetricians and Gynecologists (ACOG) guidelines

Exclusion Criteria:

* Medical or obstetric complication excluding exercise ( ACOG guideline) Major surgery or trauma in past year
* Cancer diagnosis
* Cervical incompetence
* History of ≥2 spontaneous abortions
* Multiple pregnancy
* Vaginal bleeding, placenta previa, or threatened abortion
* COPD, asthma, or chronic bronchitis
* Renal, musculoskeletal, cardiovascular, or systemic infections limiting exercise
* Polyhydramnios or oligohydramnios
* Not availability to attend to the physical exercise program

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2027-12-15 (Estimated); Study Completion 2027-12-20 (Estimated)

PRIMARY OUTCOMES:
Cardiorespiratory fitness (Vo2max) | at the 16th and 34-36th week of gestation
  The modified cycle protocol will be performed to estimate maximal oxygen uptake (VO2max), and will be used as measure of cardiorespiratory fitness.
Maternal weight gain (kg) | 34-36th week of gestation
  Maternal weight gain will be defined as the weight change from baseline measurement to the last measurement

SECONDARY OUTCOMES:
Systolic and diastolic blood pressure (mmHg) | at the 16th and 34-36th week of gestation
  Systolic and diastolic blood pressure (mmHg) will be measured after 5 minutes of rest, on 2 separate occasions (with 2 minutes between trials), with the person seated (Omron Health Care Europe B.V. Hoolddorp). The lowest value of the two trials will be selected for the analysis.
Resting heart rate (bpm) | at the 16th and 34-36th week of gestation
  Resting heart rate (bpm), will be measured after 5 minutes of rest, on 2 separate occasions (with 2 minutes between trials), with the person seated (Omron Health Care Europe B.V. Hoolddorp). The lowest value of the two trials will be selected for the analysis.
Muscle strength (kg) | at the 16th and 34-36th week of gestation
  The handgrip strength and leg press test will be used as measure of strength (upper and lower limbs)
Whole bone mineral density (g/cm2) | at the 16th to 34-36th week of gestation
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Fat free mass | at the 16th to 34-36th week of gestation
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Lean mass/fat mass ratio | at the 16th to 34-36th week of gestation
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Fat mass (kg) | at the 16th to 34-36th week of gestation
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Fat mass index (kg/m2) | at the 16th to 34-36th week of gestation
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Appendicular lean mass index (kg/m2) | at the 16th to 34-36th week of gestation
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Lean mass index (kg/m2) | at the 16th to 34-36th week of gestation
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Lean mass (kg) | at the 16th to 34-36th week of gestation
  Dual-energy X-ray absorptiometry (DXA) body composition measure
Physical activity and sedentary behaviour (in minutes) | at the 16th and 34-36th week of gestation
  Accelerometry will be used to objectively assess physical activity and sedentary time. Women will be asked to wear a tri-axial accelerometer (ActiSleep+, Pensacola, Florida, United States) for 5-7 consecutive days, starting the same day they receive the monitor (e.g. participants who receive the accelerometer on Monday, will carry the device until Tuesday of the next week).
Pittsburgh Sleep Quality Index | at the 16th and 34-36th week of gestation
  Accelerometry will be used to objectively assess physical activity and sedentary time. Women will be asked to wear a tri-axial accelerometer (ActiSleep+, Pensacola, Florida, United States) for 5-7 consecutive days, starting the same day they receive the monitor (e.g. participants who receive the accelerometer on Monday, will carry the device until Tuesday of the next week).
Quality of life (EQ-5D-5L) | at the 16th and 34-36th week of gestation
  We will use the EQ-5D-5L survey, for assessing health-related quality of life, ranging from 0 ("worst imaginable health state") to 100 ("best imaginable health state"), with higher scores representing better perceived health.
Epidemiological Studies-Depression Scale questionnaire | at the 16th and 34-36th week of gestation
  The pregnant antenatal depression levels will be assessed by the Center for Epidemiological Studies-Depression Scale questionnaire, which is validated and widely employed in pregnancy. The total score ranges from 0 to 60, with higher scores indicating more severe depressive symptoms.
Oswestry Disability Index score | at the 16th and 34-36th week of gestation
  Low-back pain will be assessed with the Spanish version of the Oswestry Disability Index (ODI) score. The final ODI score ranges from 0 to 100, where 0 represents no disability and 100 represents maximum disability.
Physical Activity index | at the 16th and 34-36th week of gestation
  Physical Activity will be assessed with the Spanish adaptation and validation of the Pregnancy Physical Activity Questionnaire (PPAQ). The scale ranges from 0 to 400+ MET·h/week, with higher scores indicating greater energy expenditure and physical activity levels.
Pain Visual Analogue Scale | at the 16th and 34-36th week of gestation
  General or specific pain intensity will also be assessed using the Pain Visual Analogue Scale (VAS), a validated self-reported measure of perceived pain intensity. The VAS consists of a 10-centimeter horizontal line anchored by "no pain" (0) and "worst imaginable pain" (10) at each end. Participants will indicate their current pain level by marking a point along the line, with higher scores representing greater pain intensity.
Cognitive Function | at the 16th and 34-36th week of gestation
  Global cognitive function will be assessed using the Montreal Cognitive Assessment (MoCA), a validated screening tool that evaluates multiple cognitive domains, including executive function, memory, attention, language, and visuospatial abilities. The total score ranges from 0 to 30, with higher scores indicating better cognitive performance.
Adherence to the Mediterranean Diet | at the 16th and 34-36th week of gestation
  Adherence to the Mediterranean dietary pattern will be assessed using the Mediterranean Diet Adherence Screener (MEDAS), a validated 14-item questionnaire designed to evaluate compliance with key components of the Mediterranean diet. Each item is scored 0 or 1, depending on whether the dietary criterion is met, yielding a total score ranging from 0 to 14, where higher scores indicate greater adherence to the Mediterranean diet.
Psychological Distress | at the 16th and 34-36th week of gestation
  The Kessler Psychological Distress Scale (K10) will be used to assess nonspecific psychological distress, including symptoms of anxiety and depression, experienced over the past four weeks. The K10 consists of 10 items, each rated on a 5-point Likert scale ranging from 1 (none of the time) to 5 (all of the time), resulting in a total score between 10 and 50. Higher scores indicate greater psychological distress.
Erythrocytes | at 34th week of gestation and at delivery
  Erythrocyte count (×10⁶ cells/µL), will be measured using an automated Coulter haematology analyser (Brand, City, Country).
Lipid profile (in mother and cord blood) | at 34th week of gestation and at delivery
  Plasma total, high-density lipoprotein and low-density lipoprotein cholesterol and triglycerides (all in mg/dL) will be assessed using an autoanalyzer.
Plasma glucose (in mother and cord blood) | at 34th week of gestation and at delivery
  Plasma glucose concentrations will be determined using the glucose oxidase enzymatic colorimetric method.
Total plasma antioxidant capacity (in mother and cord blood) | at 34th week of gestation and at delivery
  Total plasma antioxidant capacity (in maternal and cord blood) will be measured using a commercial colorimetric assay kit based on spectrophotometry, following the manufacturer's instructions. Results will be expressed in Trolox equivalents (mmol Trolox/L), where higher values indicate greater antioxidant capacity.
Antioxidant enzymes activity (in mother and cord blood) | at 34th week of gestation and at delivery
  Erythrocyte membrane catalase, glutathione peroxidase, and superoxide dismutase enzyme activities will be measured by spectrophotometry using standard biochemical assays. Results will be expressed in units per milligram of hemoglobin (U/mg Hb), where higher values indicate greater enzymatic antioxidant activity.
Pro- and anti-inflammatory signal (in mother and cord blood) | at 34th week of gestation and at delivery
  Some maternal and umbilical cord plasma pro-inflammatory and anti-inflammatory cytokines (IL-1β, IL-2, IL-6, IL-8, IL-10, IFN-γ and TNF-α, IL-1ra and TNF Srii α), some adipokines (adiponectin, adipsin, resistin, PAI-active, insulin and leptin) and myokines (irisin) will be measured by the employment of Luminex xMAP technology. Other relevant biomarkers related to bone metabolism (ACTH, DKK-1, FGF-23, Osteocalcin, OPN-Osteopontin, Osteoprotegerin, PTH and SOST) will be measured with Luminex xMAP technology. Each outcome will be reported separately, with concentrations expressed in pg/mL or ng/mL, as appropriate for the specific analyte.
Birth weight | At delivery
  Birth weight will be recorded in grams (g).
Delivery complications | At delivery
  Mode of delivery (vaginal or caesarean section) and any maternal or neonatal complications occurring during delivery will be obtained from hospital medical records and classified according to the attending obstetrician's report.
Apgar score | At delivery
  Apgar score will be evaluated at 1 and 5 minutes after delivery by trained obstetric or neonatal staff, following standard clinical procedures. Scores range from 0 to 10, with higher values indicating better neonatal condition.
Polypharmacy | At delivery and 6 and 12 months postpartum
  Polypharmacy will be defined as the concurrent use of five or more medications.
Resting energy expenditure | at the 16th and 34-36th week of gestation
  Resting energy expenditure is measured in the fasting and fed state by indirect calorimetry
Haematocrit | at 34th week of gestation and at delivery
  Haemoglobin concentration (g/dL) will be measured using an automated Coulter haematology analyser (Brand, City, Country).
Platelet count and leukocyte | at 34th week of gestation and at delivery
  Platelet count (×10³ cells/µL) and leukocyte count (×10³ cells/µL) will be measured using an automated Coulter haematology analyser (Brand, City, Country).
Mean corpuscular volume | at 34th week of gestation and at delivery
  Mean corpuscular volume (fL) will be measured using an automated Coulter haematology analyser (Brand, City, Country).
Insulin levels (in mother and cord blood) | at 34th week of gestation and at delivery
  Plasma insulin levels will be quantified by enzyme-linked immunosorbent assay (ELISA).
Glycosylated haemoglobin levels (in mother and cord blood) | at 34th week of gestation and at delivery
  Glycosylated haemoglobin (HbA1c) will be determined using the enzymatic colorimetric method.
Body length and head circumference | At delivery
  Length in centimeters (cm), and head circumference in centimeters (cm).
Hospitalization days | At delivery
  Hospitalization will be recorded as the number and duration of inpatient stays.
Cost-effectiveness analyses | At delivery and 6 and 12 months postpartum
  Cost-effectiveness analyses will be conducted based on health service utilization and associated costs extracted from the hospital database. Each outcome will be reported separately, with appropriate units (e.g., number of admissions, days hospitalized, number of medications, EQ-5D-5L index score, euros): Count (episodes, days, or medications), EQ-5D-5L index (score), and euros (€).

OTHER OUTCOMES:
Placental mitochondrial leak respiration | At delivery
  Mitochondrial oxygen (O₂) flux will be measured in placental tissue using high-resolution respirometry (Oroboros O₂k, Oroboros Instruments, Innsbruck, Austria). Tissue samples will be analyzed in fresh homogenates under controlled substrate-uncoupler-inhibitor titration (SUIT) protocols to evaluate basal, leak, and maximal respiratory states. Oxygen flux will be expressed as picomoles of O₂ consumed per second per milligram of tissue (pmol O₂·s-¹·mg-¹).
Changes to maternal, placenta and umbilical cord proteome | At delivery
  Changes in proteome will be analyzed using the Olink® proximity extension assay (PEA) technology, following the manufacturer's standardized protocol (Olink Proteomics, Uppsala, Sweden). Protein abundance will be expressed as normalized protein expression (NPX) units, where higher NPX values indicate greater relative protein concentration.

CONTACTS AND LOCATIONS:
Locations (1):
- Navarrabiomed, Hospital Universitario de Navarra (HUN) and Universidad Pública de Navarra (UPNA), Pamplona, Navarre, Spain

IPD SHARING:
Plan to Share IPD: No
This section provides details of the study plan, including how the study is designed and what the study is measuring.

REFERENCES:
- [Result] Ramirez-Velez R, Aguilar de Plata AC, Escudero MM, Echeverry I, Ortega JG, Salazar B, Rey JJ, Hormiga C, Lopez-Jaramillo P. Influence of regular aerobic exercise on endothelium-dependent vasodilation and cardiorespiratory fitness in pregnant women. J Obstet Gynaecol Res. 2011 Nov;37(11):1601-8. doi: 10.1111/j.1447-0756.2011.01582.x. Epub 2011 Jul 6. PMID 21733037
- [Result] Ramirez-Velez R, Lobelo F, Aguilar-de Plata AC, Izquierdo M, Garcia-Hermoso A. Exercise during pregnancy on maternal lipids: a secondary analysis of randomized controlled trial. BMC Pregnancy Childbirth. 2017 Nov 28;17(1):396. doi: 10.1186/s12884-017-1571-6. PMID 29179683
- [Result] Pinzon DC, Zamora K, Martinez JH, Florez-Lopez ME, de Plata AC, Mosquera M, Ramirez-Velez R. Type of delivery and gestational age is not affected by pregnant Latin-American women engaging in vigorous exercise: a secondary analysis of data from a controlled randomized trial. Rev Salud Publica (Bogota). 2012 Oct;14(5):731-43. PMID 24652353